CLINICAL TRIAL: NCT05583838
Title: Comparing the Efficacy and Safety of Optimized rhTPO Treatment Versus Eltrombopag Treatment in Previously Treated Primary Immune Thrombocytopenia Patients: A Multicenter Randomized Open-label Trial
Brief Title: A Randomized Trial Comparing Optimized rhTPO Treatment With Eltrombopag Treatment in Pre-treated ITP Pts
Acronym: TE-ITP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Xijing Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Shaanxi Provincial People's Hospital (Other); Henan Cancer Hospital (Other Government); North China University of Science and Technology (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Second Hospital of Shanxi Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Shenyang Sunshine Pharmaceutical Co., LTD. (Industry); First Affiliated Hospital of Xinjiang Medical University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Kashgar 1st People's Hospital (Other); Xi'an Central Hospital (Other); Beijing Public Health Foundation (Unknown); Yuyao People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022037
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Previously Treated Primary Immune Thrombocytopenia
Keywords: rhTPO; Eltrombopag; Pre-treated; Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Thrombopoietin; eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized rhTPO treatment (Experimental): The study in a 2:1 randomization ratio (117 subjects to rhTPO group).
  Interventions: Drug: rhTPO
- Eltrombopag treatment (Active Comparator): The study in a 2:1 randomization ratio (58 subjects to Eltrombopag group).
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: rhTPO — initial therapy: rhTPO s.c, 300 or 600U/kg daily based on baseline platelet count; maintenance therapy: rhTPO s.c, 300 ~ 600U/kg every other day depends on platelet count.
  Other Names: Recombinant human thrombopoietin; TPIAO
  Arms: Optimized rhTPO treatment
Drug: Eltrombopag — initial therapy: Eltrombopag oral, 25 or 50mg daily based on baseline platelet count; maintenance therapy: Eltrombopag oral, 25 ~ 75mg daily or every other day depends on platelet count.
  Other Names: Eltrombopag olamine
  Arms: Eltrombopag treatment

SUMMARY:
TE-ITP study: Compare the efficacy and safety of optimized rhTPO treatment versus Eltrombopag treatment in previously treated primary immune thrombocytopenia patients.

DETAILED DESCRIPTION:
A multicenter randomized open-label trial to compare the efficacy and safety of an optimized rhTPO treatment versus Eltrombopag treatment in previously treated primary immune thrombocytopenia. Total treatment duration is 6 weeks, the primary endpoint is "median time to achieve platelet count ≥50x10^9/L during 6 weeks observation".

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years old.
* Disease duration is ≥3 months, diagnosed and treated as ITP prior to screening.
* Baseline platelet count <30×10^9/L.
* Subjects treated with maintenance corticosteroids or immunosuppressive therapy must be receiving a dose that has been stable for at least 1 month.
* Informed consent has been signed.

Exclusion Criteria:

* Classified as refractory ITP.
* Subjects with any prior history of arterial or venous thrombosis, or thrombophilia in recent 1 year.
* Subjects who have previously received any platelet increasing drug such as rhTPO, thrombopoietin receptor agonist(TPO-RA), etc. within 30 days.
* Subjects who are known nonresponders to rhTPO or TPO-RA therapy.
* Subjects with positive hepatitis C virus antibody or human immunodeficiency virus(HIV) antibody, positive HBsAg and serum levels of hepatitis B virus (HBV) DNA >1000cps/ml.
* TBil or Scr> 1.5 x upper limit of normal (ULN), ALT or AST> 3.0 x ULN in recently 2 weeks.
* Subjects with any prior history of tumor.
* Female subjects who are nursing or pregnant.
* Any situation that investigate consider not suitable for pts to join the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Median time to achieve platelet count ≥50x10^9/L during 6 weeks observation | in 6 weeks treatment
  Time from the start of treatment to the first time of achieving a platelet count ≥50x10^9/L without salvage therapy during the first 6 weeks.

SECONDARY OUTCOMES:
Early response | after 1 week treatment
  Early response is defined as platelet count ≥ 30×10^9/L and at least doubling baseline at 1 week.
Initial response | after 1 month treatment
  Initial response is defined as platelet count ≥ 30×10^9/L and at least doubling baseline at 1 month.
6 weeks response | after 6 weeks treatment
  6 weeks response is defined as platelet count ≥ 30×10^9/L and at least doubling baseline at 6 weeks.
4 months response | after 4 months treatment
  4 months response is defined as platelet count ≥ 30×10^9/L and at least doubling baseline at 3 months.
Durable response | after 6 months treatment
  Durable response is defined as platelet count ≥ 30×10^9/L and at least doubling baseline at 6 months.
Time to treatment failure | in 6 weeks treatment
  Treatment failure is defined as:
  * a platelet count < 30 x 10^9/L for 4 consecutive weeks at the highest dose and schedule ; or,
  * a major bleeding event; or,
  * a change in therapy due to an intolerable side effect or bleeding symptoms (including a minor bleeding event).
Incidence of adverse events | from study start date to the end of follow-up, up to 6 months
  treatment-related adverse events.
Number of subjects with dosage under 600U/kg of rhTPO adverse events as assessed by CTCAE v5.0 | from study start date to the end of follow-up, up to 6 months
  Number of subjects with dosage under 600U/kg of rhTPO adverse events as assessed by CTCAE v5.0
Number of subjects who develop anti-rhTPO antibodies | from study start date to the end of follow-up, up to 6 months
  Number of subjects who develop anti-rhTPO antibodies
The duration time with platelet count ≥50x10^9/L | in 6 weeks treatment
  Total duration of time a subject had platelet count ≥50x10^9/L during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital,CAMS & PUMC
Locations (17):
- China (17):
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - the Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Heibei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xijing Hospital of the Fourth Military Medical University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Chinese Academy of Medical Science and Blood Disease Hospital,CAMS & PUMC, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Kashgar District 1st People's Hospital, Kashgar, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The first affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yuyao People's Hospital of Zhejiang Province, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.

REFERENCES:
- [Derived] Chen Y, Sun T, Gao D, Wang W, Zhou Z, Gao G, Wang Y, Zhou H, Song Y, Lai Y, Yan Z, Yan J, Bai J, Zhang L. Dose-optimised recombinant human thrombopoietin versus eltrombopag in patients with immune thrombocytopenia: a multicenter, randomised controlled trial (The TE-ITP Study). EClinicalMedicine. 2025 Aug 21;87:103459. doi: 10.1016/j.eclinm.2025.103459. eCollection 2025 Sep. PMID 40896456